CLINICAL TRIAL: NCT05626114
Title: A Phase IIa, Multicenter, Open-label, Single-Arm Study to Optimize Subretinal Surgical Delivery and to Evaluate Safety and Activity of Opregen in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: A Study to Optimize Subretinal Surgical Delivery and to Evaluate Safety and Activity of Opregen in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration (GAlette); Adaptive Optics (AO) Retinal Imaging Substudy in Association With Study GR44251
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR44251
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Geographic Atrophy
Keywords: Geographic Atrophy Secondary to Age-related Macular Degeneration
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OpRegen (Experimental): OpRegen dose of up to approximately 200,000 cells will be delivered into the subretinal space.
  Interventions: Biological: OpRegen

INTERVENTIONS:
Biological: OpRegen — OpRegen dose of up to approximately 200,000 cells will be delivered into the subretinal space.

SUMMARY:
This study will evaluate the success and safety of subretinal surgical delivery as well as the preliminary activity of OpRegen in participants with geographic atrophy (GA) secondary to age-related macular degeneration (AMD). All endpoints are assessed for the study eye unless otherwise indicated.

The substudy will evaluate the operational feasibility and scientific interpretability of incorporating AO retinal imaging using the EarlySight Cellularis® Discovery device. Participants who have fulfilled the eligibility requirements for the parent study and meet the substudy's eligibility criteria will have the option to participate in the substudy. The EarlySight Cellularis® Discovery device will be used only as an assessment tool and data obtained from this device will not be used to guide clinical care or influence clinical outcomes for participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to undergo a vitreoretinal surgical procedure under monitored anesthesia care
* Diagnosis of GA secondary to AMD
* Best corrected visual acuity (BCVA) score ≥ 29 letters and ≤ 60 letters in the study eye as assessed by Early Treatment Diabetic Retinopathy Study (ETDRS)
* Pseudophakic (study eye)

Exclusion Criteria:

* Pregnancy or breastfeeding
* History of cognitive impairment or dementia
* Any type of systemic disease or its treatment, in the opinion of the investigator, including any medical conditions that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical status of the participant to a significant degree or put the participant at special risk

Ocular Exclusion Criteria for Study Eye:

* Any current or history of ocular disease other than GA that may confound assessment of the macula
* History of retinal detachment
* History of vitrectomy, glaucoma-filtering surgery, or corneal transplant
* Uncontrolled glaucoma or advanced glaucoma
* Any cataract surgery or intraocular surgery within 3 months prior to subretinal surgical delivery of OpRegen
* History of other ocular or intraocular conditions that contraindicate the use of an investigational drug or may affect interpretation of the study results or may render the participant at high risk for treatment complications
* Any existing posterior segment device or implant

Substudy:

Inclusion Criteria:

- Participants must meet all of the inclusion criteria described in the parent study GR44251 and have the ability to comply with the substudy protocol

Exclusion Criteria:

* Participants who meet any exclusion criteria listed in the parent study GR44251
* Past history of seizures, or epileptic seizures due to any cause except for a single febrile seizure in childhood

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With Subretinal Surgical Delivery of OpRegen to Target Regions | 3 months post-surgery
Incidence and Severity of Procedure-related Adverse Events (AEs) at 3 Months Following Surgery | 3 months post-surgery

SECONDARY OUTCOMES:
Proportion of Participants With Qualitative Improvement in Retinal Structure, as Determined by Optical Coherence Tomography (OCT) Imaging Within 3 Months Following Surgery | 3 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (14):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Consultants Medical Group, Sacramento, California
  - West Coast Retina, San Francisco, California
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - The Retina Care Center, Baltimore, Maryland
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Cincinnati Eye Institute, Blue Ash, Ohio
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Tennessee Retina PC, Nashville, Tennessee
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Spokane Eye Clinical Research;Spokane Eye Surgery Center, Spokane, Washington
- Israel (2):
  - Hadassah MC, Jerusalem
  - Tel Aviv Sourasky MC, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Aweidah H, Matsevich C, Khaner H, Idelson M, Ejzenberg A, Reubinoff B, Banin E, Obolensky A. Survival of Neural Progenitors Derived from Human Embryonic Stem Cells Following Subretinal Transplantation in Rodents. J Ocul Pharmacol Ther. 2023 Jun;39(5):347-358. doi: 10.1089/jop.2022.0161. Epub 2023 May 4. PMID 37140896